CLINICAL TRIAL: NCT05561686
Title: Real-world Study of Pyrotinib in Neoadjuvant Therapy for HER2-positive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HunanCH-BC-001
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: HER2-positive Breast Cancer
Keywords: RWS; Pyrotinib; Neoadjuvant therapy
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum samples were collected from patients receiving pyrotinib for circulating tumor DNA (ctDNA) sequencing to calculate tumor mutation burden (TMB), and stool samples were collected to detect intestinal flora DNA (carried out according to the actual situation of the participating sites).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pyrotinib-based combination therapy: Pyrotinib, 400mg po qd, 21 days/cycle
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — This study adopted a prospective, multicenter, observational design. From October 1, 2022, 100 patients with HER2-positive breast cancer scheduled to receive neoadjuvant therapy with pyrotinib were enrolled. The treatment regimen was determined according to the patient 's condition, physician' s treatment experience, evidence-based evidence and other factors to assess the clinical benefit (pCR, ORR) and safety of different neoadjuvant therapy modalities containing pyrotinib. Exploratory analysis was performed to investigate the correlation between the level of TMB and the pCR rate of neoadjuvant therapy in HER2-positive breast cancer patients, and the effect of pyrotinib on intestinal flora.

SUMMARY:
Pyrotinib is currently being investigated in both registration studies and investigator-initiated studies in the neoadjuvant and adjuvant setting for HER2-positive breast cancer, all of which are RCTs, but randomized clinical studies have selected specific populations in defined settings, which may differ from the actual clinical setting. Given the limited real-world data on pyrotinib, real-world studies focusing on neoadjuvant therapy have not been reported. At present, we hope to collect the data of neoadjuvant therapy for HER2-positive breast cancer patients who have been prescribed pyrotinib, and explore the efficacy and safety of pyrotinib-based neoadjuvant therapy for HER2-positive early or locally advanced breast cancer patients; exploratory analysis to explore the correlation between TMB levels and pCR rate of neoadjuvant therapy in HER2-positive breast cancer patients, and the effect of pyrotinib-based neoadjuvant therapy on intestinal flora.

DETAILED DESCRIPTION:
Pyrotinib is a small molecule, irreversible, pan-ErbB receptor tyrosine kinase inhibitor that simultaneously acts on three targets, HER1, HER2, and HER4, and is stable, well tolerated, and easily penetrates the blood-brain barrier compared with macromolecular targeted drugs. In the phase II study of pyrotinib combined with capecitabine in HER2-positive breast cancer, the primary study endpoint ORR was 78.5%, and the investigator-assessed PFS reached 18.1 months with good safety; it was precisely by virtue of the phase II clinical study that the drug was preferentially approved by the State Drug Administration for marketing. During the four years of marketing, significant therapeutic effects have also been achieved in phase III clinical studies, such as the PHOEBE study and the PHENIX study; neoadjuvant treatment of patients with early and locally advanced HER2-positive breast cancer was approved for the PHEDRA study in 2022.

Pyrotinib is currently being investigated in both registration studies and investigator-initiated studies in the neoadjuvant and adjuvant setting for HER2-positive breast cancer, all of which are RCTs, but randomized clinical studies have selected specific populations in defined settings, which may differ from the actual clinical setting. Given the limited real-world data on pyrotinib, real-world studies focusing on neoadjuvant therapy have not been reported. At present, we hope to collect the data of neoadjuvant therapy for HER2-positive breast cancer patients who have been prescribed pyrotinib, and explore the efficacy and safety of pyrotinib-based neoadjuvant therapy for HER2-positive early or locally advanced breast cancer patients; exploratory analysis to explore the correlation between TMB levels and pCR rate of neoadjuvant therapy in HER2-positive breast cancer patients, and the effect of pyrotinib-based neoadjuvant therapy on intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years and ≤ 65 years
2. breast cancer meeting the following criteria: Histologically confirmed invasive breast cancer with a primary tumor > 2 cm in diameter as determined by standard assessment at the site
3. HER2 expression positive breast cancer confirmed by pathological examination, defined as an immunohistochemical (IHC) score of 3 + in > 10% of immunoreactive cells or HER2 gene amplification by in situ hybridization (ISH) results (HER2 gene signal to centromere 17 signal ratio ≥ 2.0 or HER2 gene copy number ≥ 6).
4. known hormone receptor status (ER and PgR);
5. The functional level of major organs must meet the following requirements (no blood transfusion within 2 weeks before screening, and no leukocyte-elevating or platelet-elevating drugs have been used):

1) Blood routine neutrophil (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 90 × 10^9/L; hemoglobin (Hb) ≥ 90 g/L; 2) Blood biochemistry total bilirubin (TBIL) ≤ upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; blood urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN; 3) Echocardiography left ventricular ejection fraction (LVEF) ≥ 55%; 4) 12-lead electrocardiogram Fridericia-corrected QT interval (QTcF) < 470 msec.

6. For female patients who are not postmenopausal or surgically sterile: agree to abstain from sexual activity or use an effective method of contraception during treatment and for at least 7 months after the last dose of study treatment.

7. Voluntarily join this study, sign the informed consent form, have good compliance and are willing to cooperate with the follow-up.

8. have received or plan to receive pyrotinib for neoadjuvant therapy 9. have a traceable medical history during treatment

Exclusion Criteria:

1. did not sign informed consent
2. stage IV (metastatic) breast cancer;
3. inflammatory breast cancer;
4. previous anti-tumor therapy or radiotherapy for any malignant tumor, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma and other malignant tumors;
5. Major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgical procedures;
6. serious heart disease or discomfort, including but not limited to the following diseases:

   * Confirmed history of heart failure or systolic dysfunction (LVEF < 50%);
   * High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmias (such as ventricular tachycardia) or higher grade atrioventricular block (i.e. Mobitz II second-degree atrioventricular block or third-degree atrioventricular block);
   * Angina pectoris requiring antianginal medication; -- Clinically significant valvular heart disease;
   * ECG shows transmural myocardial infarction;
   * Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
7. inability to swallow, intestinal obstruction, or other factors affecting drug administration and absorption;
8. known to be allergic to the drug components of this protocol: a history of immunodeficiency, including HIV test positive, or suffering from other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
9. pregnant and lactating women (excluding lactating women who stop breastfeeding), fertile women with positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial and within 7 months after the last dose of study drug;
10. patients who are participating in other studies
11. Have serious concomitant diseases or other conditions that would interfere with the planned treatment of concomitant diseases, or any other condition that would make the patient inappropriate for this study in the opinion of other investigators.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive breast cancer scheduled to receive pirotinib as neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Total pathologic complete response（tPCR） | Estimated 24 months
  No histological evidence of malignant tumor was found in the primary breast focus and armpit of neoadjuvant patients, or only carcinoma in situ (ypT0/is ypN0).

SECONDARY OUTCOMES:
breast pathologic complete response(bPCR) | Estimated 24 months
  No histological evidence of malignant tumor was found in the primary breast lesions of neoadjuvant patients, or only carcinoma in situ (ypt0 /is).
Objective Response Rate (ORR) | Estimated 24 months
  Ratio of CR and PR in all subjects
Adverse Events and Serious Adverse Events | From informed consent through 28 days following treatment completion
  Adverse events are described in terms of CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ying He, M.D., Study Chair — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China